CLINICAL TRIAL: NCT05091723
Title: Phase 1, Open-label Study to Assess the Pharmacokinetics and Safety of Inhaled Nezulcitinib (TD-0903) Administered in the Setting of Supplemental Oxygenation Scenarios in Healthy Participants
Brief Title: TD-0903 Pharmacokinetics Study in Healthy Participants With Supplemental Oxygenation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0196
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Acute Lung Injury (ALI) Due to Coronavirus Disease-2019 (COVID-19)
Keywords: Acute lung injury; ALI; Coronavirus Disease-2019; COVID-19; Supplemental oxygen
MeSH Terms: conditions — Acute Lung Injury; COVID-19 | interventions — nezulcitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Administration Scenario A (Experimental): Single dose of TD-0903 at Dose A on Day 1, Period 1 delivered by nasal inhalation via nebulizer device with a high-flow nasal cannula delivering supplemental oxygen
  Interventions: Drug: Nezulcitinib (TD-0903) Dose A
- Administration Scenario B (Experimental): Single dose of TD-0903 at Dose A on Day 1, Period 2 delivered by oral inhalation via nebulizer device with supplemental oxygen delivery via low-flow nasal cannula
  Interventions: Drug: Nezulcitinib (TD-0903) Dose A
- Administration Scenario C (Experimental): Single dose of TD-0903 at Dose A on Day 1, Period 3 delivered by oral inhalation via nebulizer device with supplemental oxygen delivery via high-flow nasal cannula
  Interventions: Drug: Nezulcitinib (TD-0903) Dose A
- Administration Scenario D (Experimental): Single dose of TD-0903 at Dose B on Day 1, Period 4 delivered by a route to-be-determined based on data from Scenarios A, B and C.
  Interventions: Drug: Nezulcitinib (TD-0903) Dose B

INTERVENTIONS:
Drug: Nezulcitinib (TD-0903) Dose A — TD-0903 Dose A
  Arms: Administration Scenario A; Administration Scenario B; Administration Scenario C
Drug: Nezulcitinib (TD-0903) Dose B — TD-0903 Dose B
  Arms: Administration Scenario D

SUMMARY:
This is a Phase 1 pharmacokinetic (PK) study in healthy participants to assess the plasma pharmacokinetics, safety, and tolerability of a single inhaled dose of nezulcitinib (TD-0903) with supplemental oxygenation.

DETAILED DESCRIPTION:
A Phase 1, open-label, fixed-sequence, 4-period study to evaluate the plasma PK, safety and tolerability of single inhaled doses of nezulcitinib (TD-0903) administered under different supplemental oxygenation scenarios in healthy participants.

Approximately 14 healthy adult male and female participants will receive a single inhaled dose of nezulcitinib using a nebulizer device on Day 1 of each administration period, under different supplementary oxygenations conditions.

Administration A: Dose A nezulcitinib delivered by nasal inhalation via the Aerogen Solo with a high-flow nasal cannula circuit delivering supplemental oxygen, Administration B: Dose A nezulcitinib delivered by oral inhalation via the Aerogen Solo together with the Aerogen Ultra handheld device with a low-flow nasal cannula delivering supplemental oxygen, Administration C: Dose A nezulcitinib delivered by oral inhalation via the Aerogen Solo together with the Aerogen Ultra handheld device with a high-flow nasal cannula delivering supplemental oxygen, Administration D: Nezulcitinib delivered by inhalation. Route to be determined based on data from administration A-C.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2 and weighs at least 50 kg at screening
* Medically healthy with no clinically significant medical history, physical examination, spirometry, laboratory profiles, vital signs or ECGs
* Forced expiratory volume of 1 second (FEV1) ≥80% predicted at screening and prior to dosing
* No clinically significant abnormalities in the results of laboratory
* Female subjects must be either of non-childbearing potential or if of childbearing potential, subject must not be pregnant or breastfeeding, and must agree to use a highly effective birth control method
* Male subjects must agree to use condoms to prevent potential fetal or partner exposure through seminal fluid, in addition to the use of highly effective pregnancy prevention measures with female partners of childbearing potential
* Able to understand the correct technique for the use of the nebulizer device
* Other inclusion criteria apply

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition
* Abnormal ECG measurements at screening
* Any signs of respiratory tract infection within 6 weeks of screening
* Has a current bacterial, parasitic, fungal, or viral infection; any infection requiring hospitalization or intravenous antibiotics within 6 months prior to screening
* Has any condition of the oro-laryngeal or respiratory tract
* History or presence of alcoholism or drug abuse
* Positive urine drugs of abuse test
* Positive urine or breath alcohol results
* Uses or has used tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, patches etc.) within 6 months prior to screening
* Tests positive for active COVID-19
* Additional exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Predose and at prespecified time points up to 48 hours after dosing on Day 1 of each period
  The area under the concentration time curve from time 0 extrapolated to infinity (AUC0-inf) of TD-0903
AUC0-t | Predose and at prespecified time points up to 48 hours after dosing on Day 1 of each period
  The area under the concentration time curve, from time 0 to the last observed non-zero concentration (AUC0-t) of TD-0903
Cmax | Predose and at prespecified time points up to 48 hours after dosing on Day 1 of each period
  Maximum observed concentration (Cmax) of TD-0903 in plasma

SECONDARY OUTCOMES:
Adverse Events | Day 1 through 7 following dosing on Day 1 in each of 4 Periods
  Number and severity of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.